CLINICAL TRIAL: NCT05519995
Title: The Relationship Between Sensate II Utilization and Perceived Stress in Adults
Brief Title: Sensate II Utilization and Perceived Stress in Adults
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: BioSelf Technology (Industry)
Responsible Party: Sponsor
Other Study IDs: #2022/07/14
Record Dates: First submitted 2022-08-26; First posted 2022-08-29 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Stress Disorder; Stress
Keywords: Stress; Vagus Nerve; Emotions; Sleep
MeSH Terms: conditions — Stress Disorders, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Sensate II Users: Users will be adults (18+ years of age) who have been using the Sensate II device for stress management for a minimum of 30-days or 1-month

SUMMARY:
Sensate® is A commercially marketed (FCC #: 2AS9ESEN231) stress management wellness device (BioSelf Technology; London, UK). This non-invasive wellness device is one component of a cross-modal (acoustic and aural) sensory experience designed to help an individual experience relaxation following a 10 to 30-minute session. The wellness device is paired with an in-app software program that offers infrasonic vibrations that are proprietarily synced to music or soundscapes. The wellness device is recommended in blogs, and online news articles as a possible modality for positive stress management (Bergland, 2017; Woodhall, 2018; Woolton, 2018), and anecdotal evidence from social media influencers suggest a relaxing response (Garth, 2021; Knight, 2021; Patterson, 2020). Moreover, a 2021 survey response from consumers of Sensate suggests an improvement in stress response during the COVID-19 pandemic (McDoniel & Chmelik, 2022). However, it is unknown to what extent, if any, the use of Sensate II correlated with validated measures of stress, affect, or sleep quality in adults.

DETAILED DESCRIPTION:
This study aims to assess the possible relationship between Sensate II utilization (Frequency, Duration, & Time) and perceived stress, affect, and sleep quality in adults.

1. Is there a relationship between Sensate II utilization and perceived stress
2. Is there a relationship between Sensate II utilization and postive & negative affect
3. Is there a relationship between Sensate II utilization and sleep quality. It is hypothesized that significant relationship existis between Sensate II utilization and perceived lower stress, higher postive affect, lower negative affect, and sleep quality.

References Bergland, C. (2017). Will stress-busting vagus nerve gadgetry be a game changer? Non-invasive vagus nerve stimulation reduces "fight-or-flight" stress responses. Psychology Today. http://www.psychologytoday.com/us/blog/the-athletes-way/201711/will-stress-busting-vagus-nerve-gadgetry-be-gamechanger

Garth, E. (2021). Review: Sensate stress and anxiety management. Longevity.Technology. http://longevity.technology/lifestyle/review-sensate/

Knight, S. (2021). Does the Sensate 2 do anything apart from vibrate your ribcage? http://www.makeuseof.com/sensate-review/

McDoniel, S., & Chmelik, S. (2022). A non-invasive device for stress management. https://www.researchgate.net/project/A-Non-Invasive-Wellness- Device-for-Stress-Management

Patterson, B. (2020). Sensate Meditation Device Review. http://the-gadgeteer.com/2020/07/10/sensate-meditation-device-review/

Woodhall, V. (2018). Vagus nerve: The new key to stress relief and good health. The Times. https://www.thetimes.co.uk/article/vagus-nerve-the-new-keyto- stress-relief-and-good-health-b0778h20q

Woolton, C. (2018). Wellness: Fear of flight. https://www.vogue.co.uk/article/fear-of-flying-sensate-review

ELIGIBILITY:
Inclusion Criteria:

Inclusion for this study will be adults (18+ years of age) who have been using the Sensate II device for stress management for a minimum of 30-days or one month.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults users of Sensate
Sampling Method: Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2022-08-20 (Actual); Primary Completion 2022-09-15 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress | 1-month
  Measure of perceived stress scale.
Postive Affect | 1-month
  Measure of positive Affect
Negative Affect | 1-month
  Measure of negative Affect
Sleep Quality | 1-month
  Measure of sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: Scott O McDoniel, PhD, Principal Investigator — McDoniel Holdings, LLC
Locations (1):
- BioSelf Technology, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Perceived Stress Scale, Positive / Negative Affect, & Discrete Emotions, Utilization of Sensate